CLINICAL TRIAL: NCT02315456
Title: Prospective Randomized Evaluation of Centration of Intraocular Lens With Two Laser Settings for Capsulorhexis With Femtosecond Laser
Brief Title: Evaluation of Centration of Intraocular Lens With Two Settings for Capsulorhexis With Femtosecond Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: OptiMedica Corporation (Industry)
Responsible Party: Principal Investigator, Surendra Basti, Associate Professor of Ophthalmology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1234
Record Dates: First submitted 2014-12-09; First posted 2014-12-11 (Estimated); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Capsulorhexis
Keywords: capsulorhexis; IOL centration
MeSH Terms: interventions — Capsulorhexis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Capsule centration (Other): Capsulorhexis made with capsule centration
  Interventions: Procedure: capsulorhexis
- Pupil centration (Other): Capsulorhexis made with pupil centration
  Interventions: Procedure: capsulorhexis

INTERVENTIONS:
Procedure: capsulorhexis

SUMMARY:
The study compares anatomic outcomes of Intra Ocular Lens(IOL) placement with two methods of centration of the capsulorhexis- scanned capsule centration and pupil centration. It is hypothesized that scanned capsule centration provides more uniform(25% better) overlap of capsulorhexis margin over IOL optic compared to pupil centration.

DETAILED DESCRIPTION:
50 consecutive eyes undergoing cataract surgery will be studied. 25 eyes will have scanned capsule centration and 25 will have pupil centration. Retroillumination slitlamp photographs will be taken 10-30 days after surgery with dilated pupils. The amount of capsule overlapping the IOL will be documented. The horizontal, vertical and symmetricity of overlap will be calculated.

Each group will have 20 eyes with an additional 5 eyes in each group to account for drop outs or poor quality images.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cataracts
* Same variety of IOL inserted in all eyes

Exclusion Criteria:

* Previous glaucoma or retinal surgery
* Pupil not dilating beyond 6mm
* Zonular weakness or pseudoexfoliation
* Extensive corneal scarring
* High refractive error: Myopia greater than 10D, Hyperopia greater than 5D

Ages: 45 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-08-09 (Actual); Study Completion 2016-08-09 (Actual)

PRIMARY OUTCOMES:
Overlap of the Continuous Curvilinear Capsulorhexis margin over the IOL | 10-30 days post surgery
  The horizontal and vertical overlap will be calculated. Horizontal overlap= Overlap of the temporal half versus the nasal half Vertical overlap= overlap of the superior half versus the inferior half of the IOL.
  Symmetricity of overlap= Horizontal overlap/vertical overlap

CONTACTS AND LOCATIONS:
Overall Officials: Surendra Basti, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] de Castro A, Rosales P, Marcos S. Tilt and decentration of intraocular lenses in vivo from Purkinje and Scheimpflug imaging. Validation study. J Cataract Refract Surg. 2007 Mar;33(3):418-29. doi: 10.1016/j.jcrs.2006.10.054. PMID 17321392